CLINICAL TRIAL: NCT01354834
Title: Assessment of the Clinical Efficacy of Menopur® in Intrauterine Artificial Insemination (From Partner or From Donor)
Brief Title: Assessment of the Effectiveness of Menopur in Intrauterine Insemination
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Collaborators: Ferring SAU (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Other Study IDs: FER-MEN-2003-01
Record Dates: First submitted 2011-05-16; First posted 2011-05-17 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2011-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hMG
  Interventions: Drug: hMG

INTERVENTIONS:
Drug: hMG — Patients with a condition

SUMMARY:
The purpose of this study is to assess the effectiveness of Menopur to achieve clinical pregnancy in females undergoing intrauterine insemination in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Infertile couples for over one year (primary or secondary) or infertile women (or not) with indication of PAI or DAI
* Seminal sample suitable for artificial insemination treatment according to the criterion of each centre
* Patient prescribed therapy with Menopur in artificial insemination

Exclusion Criteria:

* Contraindications to intrauterine insemination
* Contraindications to Menopur

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Females affected by infertility able to undergo intrauterine insemination
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2004-03; Primary Completion 2005-12 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 30 days

SECONDARY OUTCOMES:
Live birth rate | 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (14):
- Spain (14):
  - Investigational site, Elche, Alicante
  - Investigational site, Las Palmas, Grand Canaria
  - Investigational site, Santiago, La Coruña
  - Investigational site, Reus, Tarragona
  - Investigational site, Albacete
  - Investigational site, Alicante
  - Investigational site, Almería
  - Investigational site, Barcelona
  - Investigational site, Burgos
  - Investigational site, León
  - Investigational site, Madrid
  - Investigational site, Seville
  - Investigational site, Toldeo
  - Investigational site, Valladolid